CLINICAL TRIAL: NCT04488250
Title: Robot-Assisted Rehabilitation After HIV-Associated Stroke: Botswana
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 826195
Record Dates: First submitted 2019-04-30; First posted 2020-07-27 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS; Stroke
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Stroke

STUDY DESIGN:
Intervention Model Description: Low-to-mid functioning HIV/AIDS patients with stroke co-morbidity. Stroke survivors greater than 18 years of age with hemiplegia with and without HIV/AIDS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-to-mid functioning HIV/AIDS patients (Other): Low-to-mid functioning HIV/AIDS patients greater than 18 years of age with stroke co-morbidity.
  Interventions: Other: Robot Therapy
- Stroke survivors (Other): Stroke survivors greater than 18 years of age with hemiplegia with and without HIV/AIDS.
  Interventions: Other: Robot Therapy

INTERVENTIONS:
Other: Robot Therapy — Robot Therapy

SUMMARY:
Today, nearly 37 million people are living with HIV (PLHIV) worldwide and 30 to 40% of them will have neurologic complications leading to disability. Our long-term working hypothesis is that an effective solution for increasing rehabilitation access in Botswana and improving functional outcomes of PLHIV having experienced a stroke with or without HIV uses an affordable robot and mobile health technologies to create a cost-effective intervention strategy. For this project, we test the feasibility of affordable robot therapy.

DETAILED DESCRIPTION:
We will test the feasibility of affordable robot therapy in three Aims. In Aim 1, we will optimize for the Botswana context, an affordable technology-based robot system with four exercise stations. We will optimize a prototype of our provisionally patented robot gym system, REHAB CARES, for therapy. Optimization will include increasing cost-effectiveness, utilizing more local resources and manufacturing, and using mobile health android platforms for games and data acquisition. In Aim 2, the efficiency of the newly modified robot system compared to standard of care will be assessed using 30 patients who have experienced a stroke, with or without HIV, will be recruited from those who are being treated by Princess Marina Hospital (PMH) and living in the surrounding community. They will receive therapy using the robot gym system and receive standard of care. We will assess functional outcomes including motor impairment, function, and quality of life. The study outcomes would then inform rehabilitation practices for PLHIV with stroke, with or without HIV, and suggest that affordable technology-mediated rehabilitation can reduce their motor dysfunction and resulting long-term disability.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Stroke (at least 3 months post incident) with or without HIV, age over 18;
* medically stable (Able to tolerate therapy and given the determination as able to go through protocol by physician);
* have neurological function between 5 and 24 as defined by the NIH Stroke Scale (NIHSS);
* have no less than moderate cognitive function as defined by the International HIV-Dementia Scale
* Able to give consent.

Exclusion Criteria:

* unable to give consent;
* severely depressed (Becks Depression Inventory-Fast Screener);
* experiencing excessive pain (Visual Analog Scale (VAS) score greater than 4);
* have severe spasticity ( than 3) in muscle tone in elbow/shoulder/wrist hip/knee/ankle using the Ashworth Scale;
* have total paralysis or muscular contractures of upper or lower extremity;
* have a history of psychiatric disorder or cardiac problems;
* have a history of prior brain injury including lesions to the cerebella or brain stem;
* have open lesions on the upper or lower limbs;
* It is up to the physician to decide if a subject should be excluded due to severe drug and/or alcohol abuse or taking of medication that would impair cognitive ability.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Modified IBM Usability Satisfaction Questionnaire | At 8 Weeks
  Assess usability of the robot system with patients and therapists
Change in Baseline assessment of motor impairment | At week 8
  The Fugl-Meyer measure of motor impairment in the upper limb. Max is 66. Min 0; higher is better. up to 30 minutes to complete
Rehabilitation Capacity Questionnaire | At 0 week
  Survey for all therapists and rehab professionals - up to 1 hour; interview
Change from baseline assessment of Timed up and go | at 8 weeks
  Timed up and go - Measure gait capacity. Measured is minutes. Longer times indicate higher impairment.
Change from baseline assessment of 10 Meter Walk Test | at 8 weeks
  Measure gait distance capacity. Measured in meters. Longer distance means lower impairment.
Change from baseline assessment of # of blocks that can be grasped and moved | at 8 weeks
  Box and Block Test is a reach and grasp test - gross motor function. Measured in # of blocks. Higher number of blocks means lower impairment.
Change from baseline assessment of fine motor grasp | at 8 weeks
  Grooved Peg-Board Test is measure of fine motor grasp. Measured in times and number of pins placed. More pins placed means lower impairment.
Change from baseline assessment of stroke impact scale | at 8 weeks
  quality of life questionnaire; self-reported. The Stroke Impact Scale (SIS) assesses other dimensions of health related quality of life: emotion, communication, memory and thinking, and social role function. Higher scores means less impaired. Lower score is more impaired.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Johnson, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- Penn Medicine Rittenhouse, Philadelphia, Pennsylvania, United States
- University of Botswana, Gaborone, Botswana